CLINICAL TRIAL: NCT06086028
Title: LA-CEAL 4.0: Louisiana (LA) Community-Engagement Research Alliance (CEAL): Wearable Sensor Project
Brief Title: LA-CEAL 4.0: Wearable Sensor Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tulane University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 2023-9-19
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Results first posted 2025-10-20 (Actual); Last update posted 2025-10-20 (Actual); Status verified 2025-09

CONDITIONS: Health Care Workforce Burn Out; Stress
Keywords: Health care workforce; Burn out; Stress; Wearable sensors
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate then Delayed Arm (Experimental): The participants will receive immediate access to the data from the wearable sensor for 21 days. On day 22, all of the data from the wearable sensor will be hidden from the participant (delayed) until after the second 21-day feedback period. Wrist worn sensor: Biostrap collects biometrics such as the following: (1) sleep pattern/ quality; (2) steps, activity, calories; (3) heart rate/ HRV; (4) respiratory rate.
  Interventions: Other: Wrist worn sensor
- Delayed then Immediate Arm (Experimental): The participants begin the first 21-day feedback period with their data from the wearable sensor hidden (delayed feedback). On day 22, the wearable sensor changes to become available in real time (immediate feedback) for the second 21-day feedback period. Wrist worn sensor: Biostrap collects biometrics such as the following: (1) sleep pattern/ quality; (2) steps, activity, calories; (3) heart rate/ HRV; (4) respiratory rate.
  Interventions: Other: Wrist worn sensor

INTERVENTIONS:
Other: Wrist worn sensor — Biostrap collects biometrics such as the following: (1) sleep pattern/ quality; (2) steps, activity, calories; (3) heart rate/ HRV; (4) respiratory rate. Participants will be randomly assigned to one of two groups.

SUMMARY:
The study seeks to explore the efficacy of biofeedback collected via a wrist worn sensor in helping healthcare workers self-manage symptoms of stress and burnout.

DETAILED DESCRIPTION:
A randomized two-group cross over design will be used to test the hypothesis that using real-time biofeedback to present, interpret, and bring attention to information regarding stress levels will increase participants readiness to change in regard to addressing burnout. To test this hypothesis, the investigators will recruit 80 providers from Federally Qualified Health Centers (FQHC) partner sites to participate in a 6-week cross over design. The study includes two feedback periods: (1) 21 days of immediate information: (2) 21 days delayed information period. Participant conditions will be switched on day 22. All participants will be given a wrist worn sensor developed by Biostrap. Biostrap collects biometrics such as the following: (1) sleep pattern/ quality; (2) steps, activity, calories; (3) heart rate/ Heart Rate Variability (HRV); (4) respiratory rate. Participants will be randomly assigned to one of two groups, and either receive immediate or delayed feedback from the sensor first and will then be crossed-over to receive the opposite type of feedback. While wearing the Biostrap wrist-worn sensor, participants will be asked to complete two daily questions sent via the API. The first question seeks to determine if participants accurately understand their biometric data and will ask "how stressed are you today?" (Scale 1-10). The second question seeks to determine if participants attended to the information regarding their stress level and will ask "did you complete a self-care activity today?" (yes/no). A pre and post assessment will be given before and after completing the six-week wearable protocol. Items will include: (1) 2-item depression screener (Patient Health Questionnaire-revised) (2) 2-item anxiety screener (Generalized Anxiety Disorder Scale- revised) (3) 4-item brief resilient coping scale (4) 22-item burnout assessment (Maslach Burnout Inventory) (5) Self-care/supportive psychosocial programs utilization(e.g., I participate in an employee wellness program through my employer) (yes/no) (6) Basic demographics (e.g., age, sex, race, ethnicity, job category, years in field) (7) Familiarity and self-efficacy using wearable sensors (8) Self- report medication list (pretest only).

ELIGIBILITY:
Inclusion Criteria:

* Age >=18 years.
* Ability to understand and speak English.
* Staff at FQHC.
* Smartphone compatible with the Biostrap sensor and phone application.
* Attending work during the six week study period.

Exclusion Criteria:

* Unable or unwilling to give informed consent.
* Disclosed pregnancy at the start of the study.
* Pace maker or other device regulation heart rate/rhythm.
* Previous diagnosis of atrial fibrillation.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-05-31 (Actual); Study Completion 2024-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marie Krousel-Wood, MD, MSPH, Principal Investigator — Tulane University
Locations (1):
- Tulane School of Public Health and Tropical Medicine, New Orleans, Louisiana, United States

REFERENCES:
- [Background] Kroenke K, Spitzer RL, Williams JB. The PHQ-9: validity of a brief depression severity measure. J Gen Intern Med. 2001 Sep;16(9):606-13. doi: 10.1046/j.1525-1497.2001.016009606.x. PMID 11556941
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Sinclair VG, Wallston KA. The development and psychometric evaluation of the Brief Resilient Coping Scale. Assessment. 2004 Mar;11(1):94-101. doi: 10.1177/1073191103258144. PMID 14994958
- [Background] Maslach, C., Jackson, S. E., & Leiter, M. P. (1997). Maslach Burnout Inventory: Third edition. In C. P. Zalaquett & R. J. Wood (Eds.), Evaluating stress: A book of resources (pp. 191-218). Scarecrow Education

RESULTS

PARTICIPANT FLOW:
Groups:
- Immediate Then Delayed Arm: The participants received immediate access to the data from the wearable sensor for 21 days. On day 22, all of the data from the wearable sensor was hidden from the participant (delayed) until after the second 21-day feedback period. Wrist worn sensor: Biostrap collected biometrics such as the following: (1) sleep pattern/ quality; (2) steps, activity, calories; (3) heart rate/ HRV; (4) respiratory rate.
- Delayed Then Immediate Arm: The participants began the first 21-day feedback period with their data from the wearable sensor hidden (delayed feedback). On day 22 the wearable sensor changed to become available in real time (immediate feedback) for the second 21-day feedback period. Wrist worn sensor: Biostrap collected biometrics such as the following: (1) sleep pattern/ quality; (2) steps, activity, calories; (3) heart rate/ HRV; (4) respiratory rate.
Period: Overall Study
Arm/Group | Immediate Then Delayed Arm | Delayed Then Immediate Arm
Started | 40 | 40
Completed | 37 | 36
Not Completed | 3 | 4
Not completed — Withdrawal by Subject | 1 | 1
Not completed — Lost to Follow-up | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Immediate Then Delayed Arm: The participants will receive immediate access to the data from the wearable sensor for 21 days. On day 22 all of the data from the wearable sensor will be hidden from the participant (delayed) until after the second 21-day feedback period. Wrist worn sensor: Biostrap collects biometrics such as the following: (1) sleep pattern/ quality; (2) steps, activity, calories; (3) heart rate/ HRV; (4) respiratory rate.
- Delayed Then Immediate Arm: The participants begin the first 21-day feedback period with their data from the wearable sensor hidden (delayed feedback). On day 22 the wearable sensor changes to become available in real time (immediate feedback) for the second 21-day feedback period. Wrist worn sensor: Biostrap collects biometrics such as the following: (1) sleep pattern/ quality; (2) steps, activity, calories; (3) heart rate/ HRV; (4) respiratory rate.
- Total: Total of all reporting groups
Arm/Group | Immediate Then Delayed Arm | Delayed Then Immediate Arm | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Categorical [Count of Participants; unit: Participants] — Population: 1 participant in delayed access start arm did not respond to this question.
  Participants
    number analyzed (Participants) | 40 | 39 | 79
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 37 | 37 | 74
    >=65 years | 3 | 2 | 5
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 1 participant in delayed access start arm did not respond to this question
  years
    number analyzed (Participants) | 40 | 39 | 79
    (all) | 46.08 (12.51) | 44.92 (10.28) | 45.51 (11.40)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 1 participant in the delayed access start arm did not respond to this question
  Participants
    number analyzed (Participants) | 40 | 39 | 79
    Female | 36 | 36 | 72
    Male | 4 | 3 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: 1 participant in the delayed access start arm did not respond to this question
  Participants
    number analyzed (Participants) | 40 | 39 | 79
    American Indian or Alaska Native | 2 | 0 | 2
    Asian | 0 | 1 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 14 | 16 | 30
    White | 21 | 21 | 42
    More than one race | 1 | 0 | 1
    Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40 | 40 | 80

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Days in Concordance Comparing Immediate Information Period With Delayed Information Period
Description: The proportion of days in concordance was calculated based on responses to two questions. The first question seeks to determine if participants accurately understand their biometric data and will ask "how stressed are you today?" (Scale 1-10 a score of 6+ was coded as "high stress"). The second question seeks to determine if participants attended to the information regarding their stress level and will ask "did you complete a self-care activity today?" (yes = 1 /no = 0). Concordance was coded when participants either a) reported a high level of stress and engaged in self-care or b) when participants reported low levels of stress and did not engage in self-care. Percentage of days in concordance was calculated for both 21-day feedback periods (immediate versus delayed).
Time Frame: 6 weeks
Population: Cross-over design. 71 participants were monitored during both immediate and delayed information periods.
Measure: Mean (Standard Deviation); unit: % of days concordant
Groups:
- Immediate Information Period: Three week period during which each participant was able to view their sensor data in real time.
- Delayed Information Period: Three week period during which each participant was not able to view their sensor data in real time. They were able to view their data after the delayed information period.
Arm/Group | Immediate Information Period | Delayed Information Period
Number analyzed (Participants) | 71 | 71
% of days concordant | 0.49 (0.03) | 0.50 (0.29)

2. Secondary Outcome: Change in Burnout Score From Baseline to Follow-up (Pre/Post Sensor Data Collection)
Description: The investigators measured the change in the burnout score in all participants between baseline and 6 weeks follow-up. Maslach Burnout Inventory - Human Services Survey for Medical Personnel (MBI-HSS-MP) is a 22-item survey that covers 3 areas: Emotional Exhaustion (EE), Depersonalization (DP), and low sense of Personal Accomplishment (PA). Each subscale includes multiple questions with frequency rating choices of Never (0), A few times a year or less, Once a month or less, A few times a month, Once a week, A few times a week, or Every day (6). The total score is calculated by summing the three sub-scales and ranges from 0-132 with high scores reflecting higher symptoms of burnout and low scores reflecting fewer symptoms of burnout.
Time Frame: Baseline - 6 weeks
Population: 57 participants responded to the burnout scale on baseline and 6 weeks follow-up assessment. For this outcome measure, the burnout scale was given at baseline and at 6 weeks follow up, it was not reassessed at crossover, so the investigators didn't calculate the scale for the conditions assessed for each arm to be reported separately.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Groups:
- Baseline: Scores from baseline assessment.
- 6 Weeks Follow up: Scores from 6 weeks follow-up assessment.
Arm/Group | Baseline | 6 Weeks Follow up
Number analyzed (Participants) | 57 | 57
Change in score on a scale | 38.82 (18.48) | 35.54 (20.24)

3. Other Pre Specified Outcome: Change in Mean in Total Burnout Score of Immediate Then Delayed Arm to Delayed Then Immediate Arm
Description: The investigators measured the mean in the total burnout score of the immediate then delayed arm to the delayed then immediate arm. Maslach Burnout Inventory - Human Services Survey for Medical Personnel (MBI-HSS-MP) is a 22-item survey that covers 3 areas: Emotional Exhaustion (EE), Depersonalization (DP), and low sense of Personal Accomplishment (PA). Each subscale includes multiple questions with frequency rating choices of Never (0), A few times a year or less, Once a month or less, A few times a month, Once a week, A few times a week, or Every day (6). The total score is calculated by summing the three sub-scales and ranges from 0-132 with high scores reflecting higher symptoms of burnout and low scores reflecting fewer symptoms of burnout.
Time Frame: Baseline - 6 weeks
Population: 57 participants responded to the burnout scale on baseline and 6 weeks follow-up assessment. For this outcome measure, the total burnout score was given at baseline and at 6 weeks follow up, it was not reassessed at crossover, so the investigators didn't calculate the score for the conditions assessed for each arm to be reported separately.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Groups:
- Immediate Then Delayed Arm: The participants received immediate access to the data from the wearable sensor for 21 days. On day 22, all of the data from the wearable sensor were hidden from the participant (delayed) until after the second 21-day feedback period. Wrist worn sensor: Biostrap collected biometrics such as the following: (1) sleep pattern/ quality; (2) steps, activity, calories; (3) heart rate/ HRV; (4) respiratory rate.
Arm/Group | Immediate Then Delayed Arm | Delayed Then Immediate Arm
Number analyzed (Participants) | 32 | 25
Change in score on a scale | -2.03 (11.61) | -4.88 (16.01)

4. Other Pre Specified Outcome: Change in Mean in Total Depression Score of Immediate Then Delayed Arm to Delayed Then Immediate Arm
Description: The investigators compared the mean in total depression score of immediate then delayed arm to delayed then immediate arm. The score is a 2-item depression screener (Patient Health Questionnaire-revised). The range is from 0 to 6. The high scores reflect higher symptoms of depression, and low scores reflect fewer symptoms of depression.
Time Frame: Baseline - 6 weeks
Population: 74 participants responded to the depression questionnaire at both baseline and 6 weeks follow-up. For this outcome measure, the depression score was given at baseline and at 6 weeks follow up, it was not reassessed at crossover, so the investigators didn't calculate the score for the conditions assessed for each arm to be reported separately.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Immediate Then Delayed Arm | Delayed Then Immediate Arm
Number analyzed (Participants) | 38 | 36
Change in score on a scale | 0.08 (1.00) | -0.17 (1.18)

5. Other Pre Specified Outcome: Change in Mean in Total Anxiety Score of Immediate Then Delayed Arm to Delayed Then Immediate Arm
Description: The investigators compared the mean in total anxiety score of immediate then delayed arm to delayed then immediate arm. The score is a 2-item anxiety screener (Generalized Anxiety Disorder Scale- revised). The range is from 0 to 6. The high scores reflect higher symptoms of anxiety, and low scores reflect fewer symptoms of anxiety.
Time Frame: Baseline - 6 weeks
Population: 74 participants responded to the anxiety question at baseline and 6 weeks follow-up assessments. For this outcome measure, the total anxiety score was given at baseline and at 6 weeks follow up, it was not reassessed at crossover, so the investigators didn't calculate the score for the conditions assessed for each arm to be reported separately.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Immediate Then Delayed Arm | Delayed Then Immediate Arm
Number analyzed (Participants) | 38 | 36
Change in score on a scale | -0.05 (1.31) | -0.06 (1.49)

6. Other Pre Specified Outcome: Change in Mean in Total Resilience Score of Immediate Then Delayed Arm to Delayed Then Immediate Arm
Description: The investigators compared the mean in total resilience score of immediate then delayed arm to delayed then immediate arm. The score is a 4-item brief resilient coping scale. The range is from 4 to 20. The high scores reflect higher resilience, and low scores reflect lower resilience.
Time Frame: Baseline - 6 weeks
Population: 73 participants responded to the resilience questions on baseline and 6 weeks follow-up assessments. For this outcome measure, the total resilience score was given at baseline and at 6 weeks follow up, it was not reassessed at crossover, so the investigators didn't calculate the score for the conditions assessed for each arm to be reported separately.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Immediate Then Delayed Arm | Delayed Then Immediate Arm
Number analyzed (Participants) | 38 | 35
Change in score on a scale | 0.42 (2.54) | 0.71 (1.54)

7. Other Pre Specified Outcome: Change in Mean on Participant Sleep Score Between Immediate Information Period and Delayed Information Period
Description: The investigators measured the change in the participant sleep efficiency score in all participants between the 2 conditions to compare the difference across the conditions. Sleep efficiency score is measured via the wearable sensor. It is comprised of the following information: sleep duration (end-start), minutes in light sleep, minutes in deep sleep, stages of sleep (e.g. REM), arousal count. The range is from 0 to 100. Higher sleep efficiency scores reflect better quality sleep. Low sleep efficiency scores reflect poor quality of sleep
Time Frame: 6 weeks
Population: Cross-over design. 69 participants monitored during both immediate and delayed information periods.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Immediate Information Period | Delayed Information Period
Number analyzed (Participants) | 69 | 69
Change in score on a scale | 79.11 (13.88) | 77.21 (16.35)

8. Other Pre Specified Outcome: Change in Mean on Participant Activity Level Score Between Immediate Information Period and Delayed Information Period
Description: Activity level was measured by number of steps and distance measured by the wearable sensors. Higher scores reflect more activity while lower scores reflect less activity. An average of the daily activity level scores was calculated for each information period. Biostrap company calculated the activity score using the activity distribution over the course of a 24-hour window, emphasizing consistent physical activity of 500 steps per hour during 12 unique hours. There are no scale ranges for this activity score.
Time Frame: 6 weeks
Population: Cross-over design. 69 participants monitored in both immediate and delayed information periods.
Measure: Mean (Standard Deviation); unit: Change in score on a scale
Arm/Group | Immediate Information Period | Delayed Information Period
Number analyzed (Participants) | 69 | 69
Change in score on a scale | 62.21 (22.12) | 60.54 (23.22)

9. Other Pre Specified Outcome: Change in Respiratory Rate Between Immediate Information Period and Delayed Information Period
Description: Respiratory rate was measured as breathing rate per minute and was recorded via the wearable sensor. Higher values reflect faster breathing which is a proxy measure of stress while lower values reflect slower breathing. An average respiratory rate was calculated for each information period.
Time Frame: 6 weeks
Population: Cross-over design. 71 participants monitored in both immediate and delayed information periods.
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Immediate Information Period | Delayed Information Period
Number analyzed (Participants) | 71 | 71
Breaths per minute | 16.96 (2.00) | 16.95 (1.95)

10. Other Pre Specified Outcome: Change in Participant Heart Rate Variability (HRV) Between Immediate Information Period and Delayed Information Period
Description: HRV was calculated using root mean square of successive differences (rMSSD) using beats per minute recorded via the wearable sensor. HRV scale is 0-255. Normal scores depend on age and sex. HRV is used as a proxy measure of stress and cardiovascular health. An average HRV was calculated for each information period.
Time Frame: 6 weeks
Population: Cross-over design. 71 participants monitored in both immediate and delayed information periods.
Measure: Mean (Standard Deviation); unit: Milliseconds
Arm/Group | Immediate Information Period | Delayed Information Period
Number analyzed (Participants) | 71 | 71
Milliseconds | 32.63 (14.93) | 33.06 (15.73)

11. Other Pre Specified Outcome: Change in Participant Heart Rate Between Immediate Information Period and Delayed Information Period
Description: Heart rate is measured as beats per minute and was recorded by the wearable sensor. High values reflect faster pulse while lower values reflect lower pulse. Normal ranges for resting adult heart rate is 60 to 100. Higher heart rate is a proxy measure for stress and anxiety. An average heart rate was calculated for each information period.
Time Frame: 6 weeks
Population: Cross-over design. 71 participants monitored in both immediate and delayed information periods.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Immediate Information Period | Delayed Information Period
Number analyzed (Participants) | 71 | 71
Beats per minute | 79.00 (7.01) | 79.32 (7.75)

ADVERSE EVENTS:
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not systematically monitored/assessed.
Arm/Group | Immediate Information Period | Delayed Information Period
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT06086028/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-20): https://cdn.clinicaltrials.gov/large-docs/28/NCT06086028/SAP_001.pdf